CLINICAL TRIAL: NCT04010929
Title: Evaluation of the Efficacy of Er,Cr:YSGG Laser in Partial Pulpotomy Therapy of Permanent Immature Molar Teeth With Deep Dentin Caries
Brief Title: Efficacy of Er,Cr:YSGG Laser in Partial Pupotomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Merve Erkmen Almaz (Other)
Responsible Party: Sponsor-Investigator, Merve Erkmen Almaz, Assistant Professor, Kırıkkale University
Organization: Kırıkkale University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KirikkaleUni
Record Dates: First submitted 2019-04-19; First posted 2019-07-08 (Actual); Last update posted 2019-07-08 (Actual); Status verified 2019-07

CONDITIONS: Laser; Tooth; Pulpotomy
MeSH Terms: interventions — Pemetrexed

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Laser+MTA group (Experimental): before the MTA condensation, Er, Cr: YSGG laser was applied to the exposure area
  Interventions: Procedure: Partial pulpotomy with laser+MTA
- MTA group (Active Comparator): MTA was applied to the exposed area
  Interventions: Procedure: Partial pulpotomy with MTA

INTERVENTIONS:
Procedure: Partial pulpotomy with laser+MTA — After removing caries, laser+MTA was applied to the exposed area on the pulp following bleeding control with 5.25% NaOCl.
  Arms: Laser+MTA group
Procedure: Partial pulpotomy with MTA — After removing caries, MTA was applied to the exposed area on the pulp following bleeding control with 5.25% NaOCl.
  Arms: MTA group

SUMMARY:
The aim of this study was to compare the efficacy of partial pulpotomy treatment using MTA and Er,Cr:YSGG + MTA in permanent immature molar teeth with deep dentin caries. The study was performed in children aged between 6-15 who had at least one deep dentine caries in permanent immature molar tooth. The patients' therapies were completed in Kırıkkale University, Faculty of Dentistry, Department of Pediatric Dentisry. A total of 90 teeth (caries exposed) were included in the study. According to the treatment, the teeth were randomly divided into two groups: 1. MTA group (n=45), 2. Laser+MTA group (n=45). In the MTA group, after removing caries, MTA was applied to the exposed area on the pulp following bleeding control with 5.25% NaOCl. In the same session, the tooth was restored with resin modified glass ionomer cement and composite resin. In the laser+MTA group, the treatment procedures were the same as the MTA group, and before the MTA condensation, Er, Cr: YSGG laser was applied to the exposure area after bleeding control to provide biostimulation. Patients were called for followup appointments at 1, 3, 6 and 12 months after treatment and control radiographs were taken.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of immature molar tooth with deep dentin caries.

Exclusion Criteria:

History of any systematic disease Uncompliance with dental treatment

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 64 (Actual)
Dates: Start 2018-01-08 (Actual); Primary Completion 2019-01-14 (Actual); Study Completion 2019-01-14 (Actual)

PRIMARY OUTCOMES:
presence of spontaneous pain, percussion, palpation, mobility, presence of fistula, swelling of the mucosa, loss of lamina dura, internal or external root resorption and periapical radiolucency | First, third, sixth and twelfth month
  Presence of pathological findings were scored as 1, absence was scored as 0

CONTACTS AND LOCATIONS:
Locations (1):
- Kırıkkale University, Kırıkkale, Turkey (Türkiye)